CLINICAL TRIAL: NCT04201314
Title: Effect of InnoSlim® on Blood Sugar and Blood Lipids Regulation in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, Department of Health Diet and Industry Management, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-19062
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects take 2 starch capsules before breakfast and 3 starch capsules before dinner of similar appearance per day for 6 weeks of a stage.
  Interventions: Dietary Supplement: InnoSlim®; Dietary Supplement: Placebo
- InnoSlim® (Experimental): Subjects take 2 capsules before breakfast and 3 capsules before dinner of similar appearance per day for 6 weeks of a stage.
  Interventions: Dietary Supplement: InnoSlim®; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: InnoSlim® — Subjects take 2 capsules before breakfast and 3 capsules before dinner of similar appearance per day for 6 weeks of a stage.
Dietary Supplement: Placebo — Subjects take 2 starch capsules before breakfast and 3 starch capsules before dinner of similar appearance per day for 6 weeks of a stage.

SUMMARY:
InnoSlim® has been studied for enhancing metabolic functions whereas many lab studies have demonstrated the potential efficacy of InnoSlim® for the blood sugar and blood lipids regulation. There has been no relevant human study on InnoSlim® on blood sugar and blood lipids regulation. There have reported that 2018 estimating the total costs of diagnosed diabetes have risen to $327 billion in 2017 from $245 billion in 2012. Although pharmacological methods have been developed to treat diabetes, these treatments can be costly and are not without potential adverse effects. The development of dietary agents for the prevention of diabetes could represent a cost-effective and safe means to deal with this growing public health crisis.

DETAILED DESCRIPTION:
In this study, the investigators are investigating the effects of InnoSlim® on blood sugar and blood lipids regulation in humans. The testing sample is orally administrated to participants with pre-diabetes and hyperlipidemia humans, the efficacy parameters of blood sugar, lipid profile and other parameters, as well as adverse effects to the healthy individual, are screened during the trial, the significant difference is shown and no adverse effect reported.

ELIGIBILITY:
Inclusion Criteria:

* Participants age 20 years and above.
* Participant has provided written and dated informed consent to participate in the study.
* Participant is willing and able to comply with the study.
* Participants blood sugar (100≤ fasting blood glucose ≤ 125 mg/dL and 5.7%≤HbA1c ≤ 6.4% ) and Total cholesterol ≥200 mg/dL

Exclusion Criteria:

* Participant is participating in another clinical trial thirty days prior to enrollment.
* Participant has a significant history or current presence of treated or untreated heart disease, kidney disease, liver disease, muscle disease, bone disease, or a history of surgery.
* Participant has any medical condition or uses any medication, nutritional product, dietary supplement or program which might interfere with the conduct of the study or place the subject at risk.
* Participants lost to follow-up, non-compliance, concomitant medication.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The changes of fasting blood glucose of the subjects | 16 weeks
  A randomized-double blind, and crossover trial values change of fasting blood glucose between before to after0, 3, 6, 10, 13 & 16weeks

SECONDARY OUTCOMES:
he changes of cholesterol of the subjects | 16 weeks
  A randomized-double blind, and crossover trial values change of blood lipid between before to after0, 3, 6, 10, 13 & 16weeks
he changes of triglyceride of the subjects | 16 weeks
  A randomized-double blind, and crossover trial values change of blood lipid between before to after0, 3, 6, 10, 13 & 16weeks

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan